CLINICAL TRIAL: NCT05988697
Title: An Observational Phase II Study to Evaluate the Efficacy and Safety of Aspirin in Combination With Trametinib and Dabrafenib in Advanced Non-small Cell Lung Cancer Patients With BRAF V600E Mutation
Brief Title: Evaluate the Efficacy and Safety of Aspirin in Combination With Trametinib and Dabrafenib
Status: Not yet recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yong He, Director of Department of Respiratory Diseases, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: DATE
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: NSCLC; BRAF V600E Mutation; Advanced Cancer; Stage IIIB NSCLC; Stage IV NSCLC
Keywords: NSCLC; Asprin; Dabrafenib; Trametinib; PFS; BRAF V600E mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trametinib; dabrafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: Primary IIIB-IV BRAF V600E mutated advanced non-small cell lung cancer in a population of patients with advanced lung cancer proposed to be treated with Trametinib， Dabrafenib and Asprin
  Interventions: Drug: Combind asprin with Trametinib and Dabrafenib

INTERVENTIONS:
Drug: Combind asprin with Trametinib and Dabrafenib — Treatment drug: Dabrafenib 150 mg BID, Trametinib 2 mg QD, Aspirin 100 mg/tablet, 1 tablet/time, QD

SUMMARY:
The purpose of this study is to observe the safety and efficacy of Aspirin combined with Trametinib and Dalafenib in the treatment of advanced BRAF V600E mutated non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
lung cancer is the leading cause of morbidity and mortality in China, and non-small cell lung cancer (NSCLC) accounts for about 85% of all lung cancers. The incidence of V-Raf murine sarcoma viral oncogene homolog B1 (BRAF) mutations in NSCLC is 1.5% to 3.5%, and BRAF V600 accounts for about 30-50% of all BRAF mutations, among them, V600E mutation is the most common . NSCLC patients with BRAF V600 mutation have poor prognosis and shorter overall survival (OS). In terms of drug therapy for these patients didn't get a better clinical benefits of chemotherapy and immunotherapy, and the progression free survival (PFS) of chemotherapy is only 1.5~4.2 months . The PFS of patients with BRAF-mutated NSCLC treated with immune checkpoint inhibitors was only 3.1 to 5.3 months . In recent years, the application of targeted therapy has brought new hope for patients with lung cancer BRAF mutation. In three cohorts of the Phase II clinical trial BRF113928, the BRAF inhibitor darafenib, was demonstrated has a significant efficacy as a single agent in treated patients with BRAF V600E mutation (cohort A), combined with mitogen-activated protein kinase (MAPK) kinase (MEK) inhibitor trametinib in treated patients (cohort B), and combined with trametinib in treated patients (cohort C), respectively. Objective response rates (ORR) were 33.0%, 63.2%, and 64.0%, and PFS were 5.5, 9.7, and 14.6 months, respectively. BRF113928 research shows that Dabrafenib combined with Trametinib had good efficacy in the treatment of BRAFV600 mutant NSCLC patients, regardless of whether it was used as first-line therapy or back-line therapy, and was superior to BRAF single-agent targeted therapy. In terms of safety, the most common adverse event (AE) of Dabrafenib combined with Trametinib was fever. In cohort B and cohort C, the incidence of fever of all grades was 46% and 64%, respectively, but most of them were grade , while the incidence of grade 3-4 AE was relatively low, 2% and 11%. In general, it is safe and controllable . The main management methods for fever AE caused by Dabrafenib combined with Trametinib as follows: after the first occurrence of fever syndrome, the patient should stop taking both drugs and immediately start oral antipyretic therapy. After the fever, it is still recommended to continue the drug for 3 days before stopping the fever treatment. The selection and usage of related antipyretic drugs should be comprehensively evaluated by doctors, and the options include non-steroidal anti-inflammatory drugs, acetaminophen, and anethene. At present, the latest NCCN and CSCO both regard Dabrafenib combined with Trametinib as the preferred first-line treatment for BRAF V600E mutated advanced NSCLC patients . In March 2023, Dabrafenib combined with Trametinib entered the national medical insurance directory, reducing the economic burden of patients. However, drug resistance to targeted drugs is inevitable. Studies have shown that the resistance mechanism of BRAF/MEK inhibitors is mainly mediated by the PI3K-Akt-mtor and RAS-RAF-MEK pathways, such as cell cycle related gene changes, PI3K-AKT pathway activation, NRAS/KRAS mutations, etc. Drug resistance mechanism of Dabrafenib combined with Trametinib is complicated, there are few opportunities to use targeted drugs, also lack of clear recommendation for follow-up treatment guidelines, usually systemic treatment such as immunotherapy and chemotherapy are adopted. How to overcome the resistance mechanism, delay drug resistance, and further prolong the PFS and OS of patients of Dabrafenib combined with Trametinib still need more exploration.

Previous epidemiological studies have suggested that aspirin may reduce the incidence of certain cancers, including lung cancer. A study from the United States included 365 patients with advanced non-small cell lung cancer treated with Osimertinib, 77 of whom were taking aspirin while taking Osimertinib. The results showed that the median PFS of patients treated with aspirin was 21.3 months, which was significantly longer than the median PFS of 11.6 months of patients treated with Osimertinib alone. However, the median OS of patients treated with aspirin was lower than that of patients treated with Osimertinib alone, which was 32.3 months. Combined with aspirin could significantly reduce the risk of death of patients by 44%, suggesting that EGFR-TKI combined with aspirin could improve the patients' PFS and reduce the risk of death and bleeding events. And the same as the targeted drugs, Dabrafenib who joint Trametinib whether can combine with aspirin? How safe is it? Can the combination of aspirin with Dabrafenib and Trametinib improve the PFS and OS of patients? Aspirin has antipyretic and analgesic effects, while one of the most common adverse reactions of Dabrafenib combined with Trametinib is fever. Can the combination of Dabrafenib combined with Trametinib reduce the occurrence of adverse events of fever? At present, in the field of lung cancer, there is no literature report on aspirin combined with Dabrafenib and Trametinib in the treatment of BRAF V600E mutated advanced NSCLC. In order to solve the above problem, further improve the BRAF V600E mutations in NSCLC patients with long-term survival, we proposed the observational phase II study to evaluate the efficacy and safety of aspirin combined with Dabrafenib and Trametinib in advanced NSCLC with BRAF V600E mutation.

Primary Objectives: To determine the progression-free survival time (PFS) of aspirin combined with Dabrafenib and Trametinib;

Secondary Objectives:

A, To determine the 3 year Overall Survival (OS) in the aspirin combined with Dabrafenib and Trametinib; B, To observe the Objective Response Rate (ORR) of aspirin combined with Dabrafenib and Trametinib; C, To observe the Disease Control Rate (DCR) in aspirin combined with Dabrafenib and Trametinib; D, To observe the fever-reducing rate of aspirin combined with Dabrafenib and DabrafenibTrametinib E, To observe the risk of coronary events in patients with aspirin combined with Dabrafenib and Trametinib.

Subjects were treated with aspirin in combination with trametinib and dalafenib. The subject will be observed on the drug for 36 months, unless the subject develops tumor progression (deterioration) or a toxic reaction that is difficult to tolerate.

Treatment drug: Dabrafenib 150 mg BID, Trametinib 2 mg QD, Aspirin 100 mg/tablet, 1 tablet/time, QD.

Dabrafenib or trametinib should be interrupted or adjusted in time if a participant developed toxicity during treatment. In case of severe drug toxicity, the participant must discontinue the drug.. If the subject develops therapeutic toxicity of Asprin during the administration, the investigator shall interrupt or adjust the dose of aspirin in a timely manner. If serious drug toxicity occurs, the subject must stop taking the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Inoperable stage IIIB-IV patients with non-small cell lung cancer;
2. BRAF V600E mutation;
3. Dabrafenib and Trametinib are planned for treatment, and the survival period is expected to be more than 3 months;
4. ECOG PS 0/1;
5. The diameter of the primary lesion should be at least 1cm;
6. Previous or current aspirin treatment was allowed

Exclusion Criteria:

1. The patient is currently receiving other anticoagulant therapy;
2. The patient was previously treated with systemic anti-NSCLC;
3. The patient had other positive driver mutations, including EGFR, ALK, ROS1, MET14, RET, etc.
4. The patient had contraindications for dalafenib or trametinib and aspirin use;
5. Patients who refused follow-up visits;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is aimed at patients with advanced non-small cell lung cancer with BRAF V600E mutation in primary stage IIIB-IV. Dabrafenib and Trametinib are proposed for the treatment of advanced lung cancer
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  Progression-free survival (PFS) was calculated in 36 patients treated with aspirin combined with Dabrafenib and Trametinib
Proportion of patients with fever | C
  Refers to the proportion of patients with fever from the beginning of treatment to the end of follow-up.

SECONDARY OUTCOMES:
OS | 3 years
  3 year Overall Survival (OS) was calculated in 36 patients treated with aspirin combined with Dabrafenib and Trametinib
ORR | 3 years
  The Objective Response Rate (ORR) was calculated in 36 patients treated with aspirin combined with Dabrafenib and Trametinib. ORR will be analyzed using tests, and logistic regression methods will be used to explore other factors that influence the outcome.
DCR | 3 years
  The Disease Control Rate (DCR) was calculated in 36 patients treated with aspirin combined with Dabrafenib and Trametinib. DCR will be analyzed using tests, and logistic regression methods will be used to explore other factors that influence the outcome.
Risk of coronary events | 3 years
  Risk of coronary events was calculated in 36 patients treated with aspirin combined with Dabrafenib and TrametinibTrametinib

OTHER OUTCOMES:
Effectiveness evaluation/efficacy analysis | 3 years
  Univariate analysis of the relationship between lung cancer and treatment regimens: DFS and OS were used to compare whether there was a statistical difference (P-value less than or equal to 0.05) in the overall survival curve between the experimental and control groups by log-rank test; Multifactor analysis: PFS and OS will use a COX-proportional hazard model to estimate the hazards ratio and explore other factors that influence efficacy.
Security assessment | 3 years
  Security analysis data sets will be used for analysis. descriptive statistics, adverse events (AE), laboratory test results (blood biochemistry, liver and kidney function, coagulation and stool routine, etc.) and important vital signs (such as blood pressure) were mainly used to summarize and analyze the list.

IPD SHARING:
Plan to Share IPD: Undecided